CLINICAL TRIAL: NCT05196035
Title: A 6-month Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety and PK/PD of an age-and Body Weight-adjusted Oral Finerenone Regimen, in Addition to an ACEI or ARB, for the Treatment of Children, 6 Months to <18 Years of Age, With Chronic Kidney Disease and Proteinuria
Brief Title: A Study to Learn More About How Well the Study Treatment Finerenone Works, How Safe it is, How it Moves Into, Through, and Out of the Body, and the Effects it Has on the Body When Taken With an ACE Inhibitor or Angiotensin Receptor Blocker in Children With Chronic Kidney Disease and Proteinuria
Acronym: FIONA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19920; 2023-504884-17-00 (Registry Identifier: CTIS (EU)); 2021-002071-19 (EudraCT Number)
Record Dates: First submitted 2022-01-07; First posted 2022-01-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Chronic Kidney Disease; Proteinuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Finerenone (Kerendia, BAY94-8862) (Experimental): Participants will receive finerenone treatment.
  Interventions: Drug: Finerenone (Kerendia, BAY94-8862)
- Placebo (Placebo Comparator): Participants will receive placebo to finerenone.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone (Kerendia, BAY94-8862) — Finerenone in different doses, treatment duration will be 180±7 days
  Arms: Finerenone (Kerendia, BAY94-8862)
Drug: Placebo — Placebo to finerenone, treatment duration will be 180±7 days
  Arms: Placebo

SUMMARY:
Researchers are looking for a better way to treat children who have chronic kidney disease (CKD), which is long-term kidney disease, and proteinuria, a condition in which a person´s kidneys leak protein into the urine.

The kidneys filter waste and fluid from the blood to form urine. In children with CKD, the kidney´s filters do not work as well as they should. This can lead to accumulation of waste and fluid in the body and proteinuria. CKD can lead to other medical problems, such as high blood pressure, also known as hypertension. Vice versa, hypertension and proteinuria can also contribute to worsening of CKD. Therefore, the treatment of CKD aims to control blood pressure and proteinuria. There are treatments available for doctors to prescribe to children with CKD and hypertension and/or proteinuria. These include "angiotensin-converting enzyme inhibitors" (ACEI) and "angiotensin receptor blockers" (ARB). Both ACEI and ARB can improve kidney function by helping the renin-angiotensin-aldosterone system (RAAS) to work normally. The RAAS is a system that works with the kidneys to control blood pressure and the balance of fluid and electrolytes in the blood. In people with CKD, the RAAS is often too active, which can stop the kidneys from working properly and cause hypertension and proteinuria. However, ACEI or ARB treatment alone does not work for all patients with CKD as they only target the angiotensin part of the renin-angiotensin-aldosterone system.

The study treatment, finerenone, is expected to help control RAAS overactivation together with an ACEI or ARB.

So, the researchers in this study want to learn more about whether finerenone given in addition to either an ACEI or ARB can help their kidney function.

The main purpose of this study is to learn more about whether finerenone added to either ACEI or ARB can help reduce the amount of protein in the participants' urine more than a placebo. A placebo looks like a treatment but does not have any medicine in it. Participants will also continue to receive their other medications.

To see how the treatment work, the doctors will take samples of the participants' urine to measure their protein levels before and during taking treatment and after their last treatment. In addition, blood samples will be taken to monitor kidney function, electrolytes and the amount of finerenone in the blood as well as for other tests.

This study will include children with CKD and proteinuria aged from 6 months up to less than 18 years. The participants will take:

* either finerenone or the placebo, in addition to
* either ACEI or ARB, whichever they take as part of their normal treatment

Two visits are required up to 104 days, to check whether a child can take part in the treatment phase of the study. If participants qualify for the treatment phase, they will then undergo treatment for about 180 days. During this time, they will visit the study site at least 7 times. During these visits, the participants will:

* have their blood pressure, heart rate, temperature, height and weight measured
* have blood and urine samples taken
* have physical examinations
* have their heart examined by an electrocardiogram and echocardiography (a sonogram of the heart)
* answer questions about their medication and whether they have any adverse events , or have their parents or guardians answer
* answer questions about how they are feeling, or have their parents or guardians answer
* answer question about how they like the study medication, or have their parents or guardians answer

The doctors will keep track of any adverse events. An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

The doctors will check the participants' health about 30 days after the participants take their last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 6 months to <18 years old at the time when the informed consent/assent is signed
* Participants must have a clinical diagnosis of chronic kidney disease (CKD) at screening which is defined as

  * CKD stages 1-3 (eGFR ≥30 mL/min/1.73m^2) for children ≥1 year to <18 years of age or
  * a serum creatinine ≤ 0.40 mg/dL for infants 6 months to < 1 year of age and
  * severely increased proteinuria as defined by

    * Urinary protein-to-creatinine ratio (UPCR) of ≥ 0.50 g/g in participants ≥ 2 years with CKD stage 2 and 3 or
    * UPCR ≥ 1.0 g/g for patients < 2 years of age or ≥ 2 years of age and with CKD stage 1
* Participants must have stable kidney function between screening and D0 defined as:

  * For participants with a creatinine of > 0.8 mg/dL at screening: no increase or decrease in eGFR by ≥ 20% at D0
  * For participants with a creatinine of ≤ 0.8 mg/dL at screening: no increase or decrease in creatinine ≥ 0.15 mg/dL at D0.
* Treated with an angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) at optimized doses defined as maximally tolerable doses within the recommended dose range according to guidelines on blood pressure management, unchanged for at least 30 days prior to screening
* K+ ≤5.0 mmol/L for children ≥2 years of age at both screening and D0, and ≤5.3 mmol/L for children <2 years of age at both screening and D0

Exclusion Criteria:

* Planned urological surgery expected to influence renal function
* Children with hemolytic uremic syndrome (HUS) diagnosed ≤6 months prior to screening
* Patients with nephrotic syndrome receiving albumin infusions within the last 6 months prior to screening
* Patients who are candidates for renal transplantation, i.e., a kidney transplantation scheduled within the study time frame
* Renal allograft in place
* Bilateral renal artery stenosis
* Acute kidney injury requiring dialysis within 6 months prior to screening
* Systemic hypertension stage 2 in children ≥1 year of age defined according to guidelines on blood pressure management at screening or randomization
* Systolic blood pressure (SBP) above 110 mmHg in infants 6 months to <1 year of age at screening or randomization
* Systemic hypotension defined as a systolic blood pressure below the 5th percentile for age, sex and height at either screening or randomization but no lower than 80 mmHg (although for some participants the 5th percentile of SBP is < 80 mmHg they must be excluded if their SBP is <80 mmHg)
* Participants with immune-mediated CKD using rituximab, cyclophosphamide, abatacept, or high-dose glucocorticoids, within <6 months prior to screening

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 219 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Percent change in Urinary protein-to-creatinine ratio (UPCR) reduction from baseline to day 180+/-7 | From baseline to day 180+/-7
  Percent change from baseline to day 180±7 in UPCR will be calculated.

SECONDARY OUTCOMES:
Number participants with treatment emergent adverse events (TEAEs） | From the start of study intervention to last study intervention + 3 days (up to 190 days)
  Below sub-categories will be considered:
  1. Serious Treatment Emergent Adverse Events (TEAEs)
  2. TEAEs and serious TEAEs leading to discontinuation of treatment
  3. Study drug related TEAEs and serious TEAEs
  4. TEAEs categorized by severity (mild, moderate, severe)
  5. TEAEs by maximum intensity
  6. Number of participants hospitalized with hyperkalemia,
  7. Number of participants discontinuing due to hyperkalemia,
  8. Number of participants with hospitalization for worsening of renal function
  9. Number of participants discontinuing due to worsening of renal function
Change in serum potassium levels from baseline to day 180±7 | From baseline to day 180±7
Change in serum creatinine from baseline to day 180±7 | From baseline to day 180±7
Change in eGFR from baseline to day 180±7 | From baseline to day 180±7
  Estimated glomerular filtration rate (eGFR)
Change in systolic blood pressure from baseline to day 180±7 | From baseline to day 180±7
UPCR reduction of at least 30% from baseline to day 180+/-7 | From baseline to day 180±7
  Proportion of participants at day 180+/-7 with a >=30% reduction in PUCR compared to baseline
Change in UACR from baseline to day 180±7 | From baseline to day 180±7
  Urinary albumin-to-creatinine ratio (UACR)
Pharmacokinetics (PK) finerenone Cmax, md | Pre-dose, post-dose (1.5-5 hours after intake of intervention), up to day 180±7
  Maximum observed finerenone concentration in plasma after multiple doses.
Pharmacokinetics (PK) finerenone AUCτ,md | Pre-dose, post-dose (1.5-5 hours after intake of intervention), up to day 180±7
  Area under the curve for finerenone concentration in plasma after multiple doses.
Taste and texture questionnaire of the pediatric formulation | On day 30±3 and day 180±7

CONTACTS AND LOCATIONS:
Locations (154):
- United States (18):
  - Phoenix Children's Hospital | Main - Transplant Department, Phoenix, Arizona
  - Cedars-Sinai Medical Center - Nephrology, Los Angeles, California
  - Lucille Packard Children's Hospital Stanford - Pediatric Nephrology, Palo Alto, California
  - Rady Children's Hospital San Diego - Cardiology, San Diego, California
  - Children's National Hospital - Nephrology, Washington D.C., District of Columbia
  - Memorial Transplant Institute - Pediatric Nephrology, Hollywood, Florida
  - Emory University Hospital/Children's Healthcare of Atlanta - Nephrology, Atlanta, Georgia
  - University of Iowa Health Care Medical Center - Nephrology, Iowa City, Iowa
  - The Charlotte R. Bloomberg Children's Center Building - Nephrology, Baltimore, Maryland
  - Boston Children's Hospital - Main Campus - Nephrology, Boston, Massachusetts
  - Children's Mercy Hospital Kansas City - Nephrology, Kansas City, Missouri
  - Cincinnati Children's Hospital Medical Center | Division of Nephrology and Hypertension, Cincinnati, Ohio
  - Cleveland Clinic | Pediatric Nephrology, Cleveland, Ohio
  - OHSU Doernbecher Children's Hospital - Neurology, Portland, Oregon
  - Children's Hospital of Philadelphia - Nephrology, Philadelphia, Pennsylvania
  - Univ of Texas Health Science Center | Nephrology Res Dept, San Antonio, Texas
  - Eccles Primary Children's Outpatient Services - Nephrology, Salt Lake City, Utah
  - Seattle Children's Hospital - Nephrology, Seattle, Washington
- Argentina (6):
  - Instituto Universitario Hospital Italiano de Buenos Aires | Hospital Italiano de Buenos Aires - Neurology Department, Ciudad Autonoma de Buenos Aire, Ciudad Auton. de Buenos Aires
  - Hospital General de Ninos Ricardo Gutierrez | Pediatric Nephrology Department, Ciudad Autonoma de Buenos Aire, Ciudad Auton. de Buenos Aires
  - Centro de Rehabilitacion Cardiovascular | San Luis, Argentina, San Luis, San Luis Province
  - Clinica de Nefrologia, Urologia y Enfermedades Cardiovascualares | Santa Fe, Argentina, Santa Fe, Santa Fe Province
  - Hospital de Pediatría Juan P. Garrahan, Buenos Aires
  - Hospital General de Ninos Pedro de Elizalde | Nephrology Department, Buenos Aires
- Australia (3):
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Monash Children's Hospital, Clayton, Victoria
  - Royal Children's Hospital Melbourne, Parkville, Victoria
- Austria (4):
  - Medizinische Univ Graz | Kinder & Jugendheilkunde, Graz, Styria
  - Kepler Universitätsklinikum Campus IV, Innsbruck, Tyrol
  - Uniklinikum Salzburg - Landeskrankenhaus, Vienna, Vienna
  - AKH Wien | Kinder & Jugendheilkunde, Kindernephrologie, Vienna, Vorarlberg
- Belgium (5):
  - Huderf / Ukzkf, Bruxelles - Brussel
  - CU Saint-Luc/UZ St-Luc, Bruxelles - Brussel
  - UZ Gent, Ghent
  - UZ Gasthuisberg - Pediatric Nephrology, Leuven
  - CHC Montlégia - Pediatrics, Liège
- Brazil (6):
  - Instituto da Crianca e do Adolescente, São Paulo, Ceará
  - Hospital Pequeno Principe, Curitiba, Estado de Bahia
  - Hospital PUC-Campinas | Centro de Pesquisa Clínica Sao Lucas, São Paulo, Estado de Bahia
  - Hospital Infantil Sabará - Instituto PENSI - Pesquisa e Ensino em Saúde Infantil, São Paulo, Minas Gerais
  - Hosp Clínicas Facult. Med. de Ribeirão Preto / USP, Ribeirão Preto/SP, Rio de Janeiro
  - Santa Casa de Misericórdia de Belo Horizonte, São Paulo, Rio Grande do Sul
- Bulgaria (3):
  - UMHAT Sveti Georgi, Plovdiv
  - SHATPD "Prof. Ivan Mitev", Sofia
  - MHAT prof. Stoyan Kirkovitch AD, Stara Zagora
- Canada (3):
  - Alberta Children's Hospital - Nephrology Clinic, Calgary, Alberta
  - McMaster Children's Hospital, Hamilton, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- Czechia (2):
  - Všeobecná fakultní nemocnice v Praze, Prague
  - Fakultní nemocnice Motol a Homolka, Pracovište MOTOL, Prague
- Denmark (3):
  - Aarhus Universitetshospital - Børn og Unge, Århus N
  - Rigshospitalet - Børn og Unge, Copenhagen
  - Odense Universitetshospital - HC Andersen Børne og Ungehospital, Odense C
- Finland (3):
  - HUS-Yhtymä, Helsingin yliopistollinen sairaala (HUS) - Uusi lastensairaala, nefrologia, Helsinki
  - Tampere University Hospital, Tampereen yliopistollinen sairaala (TAYS) - Lasten lääketutkimuskeskus PeeTU, Tampere
  - Turun yliopistollinen keskussairaala, Turku
- France (6):
  - CHU bordeaux - Hopital Pellegrin, Bordeaux
  - CHU de Lyon - Hopital Femme Mère Enfant, Bron
  - Hopital Arnaud de Villeneuve CHU Montpellier, Montpellier
  - Hopital Robert Debre, Paris
  - CHU Strasbourg - Hopital Hautepierre, Strasbourg
  - Hôpital des Enfants, Toulouse
- Germany (7):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Medizinische Hochschule Hannover (MHH), Hanover, Lower Saxony
  - Kindernierenzentrum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Charité / Pädiatrie, Berlin
  - Universitätsklinikum Hamburg Eppendorf (UKE), Hamburg
- Greece (5):
  - Children's Hospital of Athens P&A Kyriakou - Pediatric Nephrology Department, Athens
  - Children's Hospital of Athens Agia Sofia - Pediatric Nephrology Department, Athens
  - University General Hospital of Heraklion - Department of Paediatrics, Heraklion
  - University General Hospital Of Ioannina-Child Health Sector, Ioannina
  - Ippokratio General Hospital Of Thessaloniki-Pediatric Nephrology Unit, 3rd Department of Paediatrics, Thessaloniki
- Hungary (4):
  - Semmelweis University, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - SZTE ÁOK Szent Györgyi Albert Klinikai Kozpont, Szeged
- India (6):
  - Institute of Kidney Diseases and Research Center Gujarat University of Transplantation Sciences, Ahmedabad, Gujarat
  - Mavani Kidney Care, Ahmedabad, Gujarat
  - St. John's National Academy of Health Sciences, Bengaluru, Karnataka
  - All India Institute of Medical Sciences (AIIMS) - New Delhi, Delhi, National Capital Territory of Delhi
  - NRS Medical college, Kolkata, West Bengal
  - Post Graduate Institute of Medical Education and Research, Chandigarh
- Israel (5):
  - Clalit Health | Soroka Medical Center - Internal Medicine Department, Beersheba
  - Wilf Children's Hospital Shaare Zedek Medical Center, Jerusalem
  - Health Corporation of Galilee Medical Center, Nahariya
  - Clalit Health Services Schneider Children's Medical Center, Petah Tikva
  - Dana-Dwek Children's Hospital, Tel Aviv
- Italy (6):
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS_Policlinico Sant'Orsola - Pediatria, Bologna, Emilia-Romagna
  - Ospedale Pediatrico Bambino Gesù - Nefrologia, Rome, Lazio
  - IRCCS Istituto Giannina Gaslini - Nefrologia e Trapianto Rene, Genoa, Liguria
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Nefrologia e Dialisi Pediatrica, Trapianti di Rene, Milan, Lombardy
  - Azienda Ospedaliera Universitaria Meyer IRCCS - Nefrologia e Dialisi, Florence
  - A.O.U. Città della Salute e della Scienza di Torino_Regina Margherita - Nefrologia Pediatrica, Torino
- Lithuania (2):
  - Hospital of LT University of Health Sciences Kaunas Clinics, Kaunas
  - Vilnius University Hospital Santaros Klinikos Children's Hospital Paediatrics Centre, Vilnius
- Malaysia (5):
  - Hospital Tunku Azizah, Wilayah Persekutuan, Kuala Lumpur
  - Hospital Tuanku Ja'afar, Seremban, Negeri Sembilan
  - Hospital Selayang, Shah Alam, Selangor
  - Sunway Medical Centre, Subang Jaya, Selangor
  - Hospital Universiti Sains Malaysia, Kelantan
- Mexico (6):
  - Sitio Alfredo Chew Wong | Aguascalientes, Mexico, Aguascalientes, Agguascalientes
  - Instituto Veracruzano en Investigación Clinica SC, Mexico City, Mexico City
  - Hospital Infantil de México "Dr. Federico Gómez", México D.F., Mexico City
  - Instituto Nacional de Pediatría, México, D.F., Mexico City
  - Hospital Universitrio Dr. José Eleuterio González. Servicio de Oncologia, Nuevo León, Monterrey
  - Hospital Regional de Alta Especialidad Ixtapaluca, Ixtapaluca, State of Mexico
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - University Medical Center Utrecht, Utrecht
- Poland (6):
  - Uniwersytecki Dzieciecy Szpital Kliniczny im. L. Zamenhofa, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw
  - Uniwersytecki Szpital Kliniczny UM we Wroclawiu, Wroclaw
- Portugal (2):
  - Hospital Pediátrico de Coimbra I ULS Coimbra, Coimbra
  - Unidade Local de Saúde de Santo António, E.P.E, Porto
- Wits Vaccines & Infectious Diseases Analytics (VIDA) Research Unit, Soweto, Gauteng, South Africa
- South Korea (5):
  - Kyungpook National University Hospital, Daegu, Daegu Gwang''yeogsi
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Korea University Guro Hospital, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
- Spain (6):
  - Hospital Universitari Vall D Hebron | Nefrologia pediatrica, Barcelona
  - Hospital Sant Joan De Deu Barcelona | Nefrologia pediatrica, Barcelona
  - Hospital Universitario 12 De Octubre | Nefrologia pediatrica, Madrid
  - Hospital Universitario La Paz | Nefrologia pediatrica, Madrid
  - Hospital Universitario Regional De Malaga | Nefrologia pediatrica, Málaga
  - Hospital Universitario Virgen Del Rocio S.L. | Nefrologia pediatrica, Seville
- Sweden (3):
  - Skånes Universitetssjukhus Lund - Barnnefroenheten, Lund
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala
- Switzerland (3):
  - Universitäts-Kinderspital UKBB, Basel, Canton of Basel-City
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - Hopital des Enfants HUG, Geneva
- Taiwan (6):
  - National Cheng Kung University Hospital, Tainan, TNN
  - Chang Gung Memorial Hospital (CGMH) - Kaohsiung Branch, Guishan
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (8):
  - Cukurova Univ. Tip. Fak. Balcali Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Baskent Universitesi Tip Fakultesi Hastanesi, Ankara
  - Gazi Universitesi Tip Fakultesi, Ankara
  - T.C. Saglik Bakanligi Ankara Bilkent Sehir Hastanesi Noroloji ve Ortopedi Hastanesi Noroloji Bolumu, Ankara
  - Istanbul Faculty of Medicine, Department of Internal Medicine, Department of Pediatrics, Istanbul
  - Istanbul Universitesi Cerrahpasa - Cocuk Nefrolojisi, Istanbul
  - Marmara University Medical Faculty | Pediatric Nephrology, Istanbul
- United Kingdom (4):
  - Great Ormond Street Hospital for Children NHS Foundation Trust | Great Ormond Street Hospital - Clinical Research Facility, London, Greater London
  - Manchester University NHS Foundation Trust | Royal Manchester Children's Hospital - Clinical Research Facility, Manchester, Greater Manchester
  - Nottingham University Hospitals NHS Trust | Queens Medical Centre - Childrens Clinical Research Facility, Nottingham, Nottinghamshire
  - NHS Greater Glasgow and Clyde | Royal Hospital for Children - Glasgow Clinical Research Facility, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Schaefer F, Montini G, Kang HG, Walle JV, Zaritsky J, Schreuder MF, Litwin M, Scalise A, Scott H, Potts J, Iveli P, Breitenstein S, Warady BA. Investigating the use of finerenone in children with chronic kidney disease and proteinuria: design of the FIONA and open-label extension studies. Trials. 2024 Mar 21;25(1):203. doi: 10.1186/s13063-024-08021-z. PMID 38509517